CLINICAL TRIAL: NCT06234384
Title: Foundation for Sarcoidosis Research Advanced Cures Registry (FSR-SARC Registry)
Status: Recruiting | Type: Observational
Sponsor: Foundation for Sarcoidosis Research (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00008556
Record Dates: First submitted 2024-01-16; First posted 2024-01-31 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Sarcoidosis diagnosis — Participants have been diagnosed with sarcoidosis.

SUMMARY:
The goal of the study is to create a longitudinal record of patient reported outcomes for people living with sarcoidosis that maintains privacy. Patients report on the following: demographics, disease symptoms, diagnostic journey, provider experience, disease treatment, and burden of disease. Patients can also link their Electronic Health Records (EHR). The goal is to create a natural history of sarcoidosis, support research, and better understand the needs of the sarcoidosis community.

DETAILED DESCRIPTION:
Participants review a document, Understanding Your Participation, and check boxes on the Participant Informed Consent document that confirms they understand the risks/benefits of participation (or Assent if the patient is a minor age 7-18), they create an online account, and then are asked to complete the baseline survey questionnaire. Participants confirm they understand that their participation is completely voluntary, that their identifying information will be secured and encrypted, their private health information will be stored separately in a secure database. Their private information will never be shared with other people, unless its required by law. The registry may share de-identified information with researchers and other databases. Their personal information will be protected and not shared. They may choose to stop their participation at any time by contacting FSR. They are not required to fill out all the questions and can leave any unanswered. They will be contacted by the registry once a year to update or correct their health information. They can choose to be contacted by FSR if a study becomes available that they may wish to know more about.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. Consent
3. Sarcoidosi diagnosis -

Exclusion Criteria:

NONE

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any adult or child (with a parent or legal guardian's assent) who has been given the diagnosis of sarcoidosis (including juvenile sarcoidosis or Blau Syndrome), and who are able to understand the consent form explaining the risks and benefits of participation.
Sampling Method: Non-Probability Sample
Enrollment: 6833 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2033-06 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Completed participation in baseline survey | If a survey question is completely blank, a query can be sent to request the subject to complete the section. Subjects will be contacted only twice to attempt to resolve an issue. The timeframe from time to event outcome shall not exceed 6 months.
  Baseline survey completion

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation For Sarcoidosis Research, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
All patient data is de-identified, researchers can request access to de-identified data only.